CLINICAL TRIAL: NCT05667220
Title: Efficacy of Combination Therapy With Sitagliptin and Beidougen Capsule in Chinese Patients With Type 2 Diabetes
Brief Title: Sitagliptin in Combination With Beidougen Capsule for Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Beijing Chao Yang Hospital, Beijing Chao Yang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-Sitagliptin-Beidougen
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin monotherapy group (Group A) (Active Comparator)
  Interventions: Drug: Sitagliptin
- Sitagliptin combined with Beidougen capsule treatment group (Group B) (Experimental)
  Interventions: Drug: Sitagliptin combined with Beidougen capsule

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin monotherapy group (Group A): 20 eligible patients were planned to be included and given Sitagliptin 100 mg Qd orally; the treatment period was 1 week.
  Arms: Sitagliptin monotherapy group (Group A)
Drug: Sitagliptin combined with Beidougen capsule — Sitagliptin combined with Beidougen capsule treatment group (Group B): 20 eligible patients were planned to be included and given sitagliptin 100mg Qd orally combined with Beidougen capsule 60mg Tid orally. The treatment period was 1 week.
  Arms: Sitagliptin combined with Beidougen capsule treatment group (Group B)

SUMMARY:
The study was an interventional non-randomized controlled study and was divided into a Sitagliptin monotherapy (100 mg Qd) group and a Sitagliptin (100mg Qd)+Beidougen capsule (60mg Tid) combination treatment group for one week.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years with a first diagnosis of type 2 diabetes
* Diagnostic criteria HbA1c ≥ 7%

Exclusion Criteria:

* The positive of diabetes antibodies
* Anti-diabetic drugs therapy before participation
* Pancreatitis
* Coronary artery disease
* Liver function impairment
* Renal function impairment
* History of intestinal surgery
* Chronic hypoxic diseases (emphysema and cor pulmonale)
* Infectious disease
* Hematological disease
* Systemic inflammatory disease
* Cancer
* Pregnant
* Ingesting agents known to influence glucose or lipid metabolism
* Any antibiotics or probiotics in the past three months prior to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose change | Changes in fasting blood glucose from baseline to 1 week treatment
  Fasting blood glucose (FBG) levels (mmol/L) were analyzed by an autoanalyzer (Hitachi 747, Roche Diagnostics, Germany) at the Central Chemistry Laboratory of Beijing Chaoyang Hospital affiliated with Capital Medical University.

SECONDARY OUTCOMES:
Serum GLP-1 change | Changes in serum GLP-1 from baseline to 1 week treatment
  The serum active GLP-1 contents were measured using an active GLP-1 assay kit (EZGLPHS-35K, Millipore) according to the specification.
Fecal DPP4 activity change | Changes in fecal DPP4 activity from baseline to 1 week treatment
  For measurement of fecal DPP4 activity, 60 mg feces were homogenized in RIPA lysis buffer (with final concentration at 1 mg/mL) was added to 50 mM sodium phosphate buffer (pH = 7.4, OD600 = 0.5), and the reaction was started by the addition of 250 μM H-A-pNA. After incubation for 30 min at 37 °C, the absorbance was measured at 405 nm.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Wang, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China